CLINICAL TRIAL: NCT02204930
Title: A Multi-centre, Open-label, Uncontrolled, First-in-Human Study to Evaluate the Safety and Tolerability and Explore the Efficacy of PeproStat in Gelita-Spon® Gelatin Sponge in Subjects Undergoing Open Liver Resection Surgery
Brief Title: PeproStat Haemostat Study in Subjects Undergoing Liver Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haemostatix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HX-01-UK; 2013-001993-10 (EudraCT Number)
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Hemorrhage
Keywords: Haemostat; Liver surgery; Primary liver cancer; Metastatic liver cancer; Benign liver disease such as adenoma; Hepatitis-related or alcoholic-related liver cirrhosis; Living donation for liver transplant
MeSH Terms: conditions — Hemorrhage; Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Haemostat (Experimental): PeproStat
  Interventions: Drug: PeproStat

INTERVENTIONS:
Drug: PeproStat — A solution of PeproStat containing up to 9.25mg protein soaked immediately prior to use onto a Gelita-Spon® gelatin sponge.

SUMMARY:
The purpose of this First in Man study is to evaluate the safety and tolerability, as well as to explore efficacy of PeproStat, a new peptide based coagulant (haemostat), when used in patients undergoing open liver resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Are able and willing to provide written informed consent to participate in this study, confirmed by signing the informed consent documents
* Adult males and females ≥18 years of age
* Female subjects must be post-menopausal. Post-menopausal status is defined as any of the following: natural menopause with menses >1 year ago; radiation induced oophorectomy with last menses >1 year ago; chemotherapy induced menopause with 1 year interval since last menses
* Willing and able to comply with all protocol requirements including follow-up
* Subject must have a haemoglobin ≥ 9.0 g/dL at screening
* Subject must have a platelet count ≥ 100,000/mm3 at screening
* Subject is undergoing a planned open liver resection
* Male subjects must be willing and able to use adequate contraception from enrollment through to the 30 day follow-up visit
* During the surgery, the subject presents an identified target bleeding site (TBS) with oozing, mild or moderate bleeding, which conventional surgical techniques are insufficient to control and would otherwise be a candidate for standard haemostats
* During the surgery, subject presents no intraoperative complications, other than bleeding, that may interfere with study assessments as judged by the investigator

Exclusion Criteria:

* Subject is undergoing emergency surgical procedure
* Recipient of a liver transplant
* Females of child-bearing potential
* Active infection at the time of the liver resection
* International Normalized Ratio (INR) > 2.0 or APTT ratio > 2.0 at screening
* Fibrinogen level < 1.5g/L at screening
* History of thromboembolic disease and/or thrombophilia
* Any other disease or condition that may affect normal blood clotting, for example thrombocytopenia, as judged by the investigator
* A known history of anaphylaxis or allergic reaction to human albumin, PEGylated proteins, yeast or moulds, porcine products or other components in the IMP
* Participation in another investigational drug or device research study within 30 days before and after enrolment in the current study
* Current known or suspected alcohol and/or drug abuse or dependence at the time of screening
* Any concurrent medical, surgical, or psychiatric condition that may, in the investigator's opinion, affect the subject's willingness or ability to meet all study requirements during the study duration
* During the surgery, subject presents severe bleeding where use of a topical haemostat would be inappropriate
* Subject is taking any prohibited medications
* BMI at screening of ≥35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety of PeproStat | within 30 days after surgery and study treatment
  Incidence, severity, and relatedness of adverse events (AEs) and adverse drug reactions (ADRs).

SECONDARY OUTCOMES:
Assessment of efficacy of PeproStat in achieving haemostasis in open liver resection surgery | During surgery
  Percentages of subjects who achieve haemostasis within 3, 5, 7 and 10 minutes following application for the first five subjects and at 1, 3, 5, 7 & 10 minutes following application in subsequent subjects.
Assessment of efficacy of PeproStat in achieving haemostasis in open liver resection surgery | During surgery
  Mean time to haemostasis.
Assessment of efficacy of PeproStat in achieving haemostasis in open liver resection surgery | During surgery
  Percentage of subjects who do not achieve haemostasis within 10 minutes.
Assessment of efficacy of PeproStat in achieving haemostasis in open liver resection surgery | During surgery
  Administered dose of PeproStat determined by number of sponges administered to a single bleeding site.

OTHER OUTCOMES:
Exploratory Immunogenicity | within 30 days after surgery and study treatment
  Immunogenicity to be investigated using a specific antibody test which has been established but not yet validated.

CONTACTS AND LOCATIONS:
Overall Officials: D Mirza, MBBS, MS, FRCS, Principal Investigator — The Queen Elizabeth Hospital
Locations (4):
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrooke's University Hospital, Cambridge
  - Kings University Hospital, London
  - Derriford Hospital, Plymouth